CLINICAL TRIAL: NCT06125704
Title: The Time to Move Randomized Crossover Trial
Brief Title: Time to Move in Pregnancy Hyperglycemia
Acronym: TtM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Samantha Ehrlich, Assocaite Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: TtM
Record Dates: First submitted 2023-10-30; First posted 2023-11-09 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: GDM; Physical Activity; Hyperglycemia; Glucose Intolerance; Circadian Rhythm; Exercise
MeSH Terms: conditions — Motor Activity; Hyperglycemia; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning physical activity first (Other): Randomized to complete 30 minute of moderate intensity walking or stepping in the morning (i.e., between 5am-9am, within 30-40 minutes of starting breakfast) on days 4 and 5, and 30 minute of moderate intensity walking or stepping in the late afternoon/evening (between 4pm-8pm, within 30-40 minutes of dinner) on days 9 and 10.
  Interventions: Behavioral: Moderate intensity walking or stepping
- Afternoon/evening physical activity first (Other): Randomized to complete 30 minute of moderate intensity walking or stepping in the late afternoon/evening (between 4pm-8pm, within 30-40 minutes of dinner) on days 4 and 5, and 30 minute of moderate intensity walking or stepping in the morning (i.e., between 5am-9am, within 30-40 minutes of starting breakfast) on days 9 and 10.
  Interventions: Behavioral: Moderate intensity walking or stepping

INTERVENTIONS:
Behavioral: Moderate intensity walking or stepping — 30 minutes of moderate intensity walking or stepping (i.e., at a pace of approximately 100 steps per minute), varied by time of day it is performed: morning (i.e., between 5am-9am, within 30-40 minutes of starting breakfast) versus late afternoon/evening (i.e., between 4pm-8pm, within 30-40 minutes of dinner).

SUMMARY:
This randomized controlled crossover trial of 36 pregnant individuals with gestational diabetes (GDM) or gestational glucose intolerance (GGI) will:

1. Determine the effects of physical activity (PA) timing, specifically 30 minutes of moderate intensity walking or stepping in the morning (between 5am-9am, within 30-40 minutes of starting breakfast), versus late afternoon/evening (between 4pm-8pm, within 30-40 minutes of dinner) on glucose across the 24-hour cycle.
2. Explore the potential effects of the timing of PA on sleep and mood state.

DETAILED DESCRIPTION:
Research participants will:

1. Exercise according to a schedule provided by the study for an 11-day period. They will complete either no exercise or 30 minutes of walking/stepping (e.g., stepping in place or around the house when walking outside is not an option or not an attractive option) on specifically assigned days, at specifically assigned times of day.
2. Wear a masked Dexcom G6 continuous glucose monitor (CGM) or unmasked Dexcom G7 CGM for the 11-day study period.
3. Wear a masked physical activity (PA) monitor watch (ActiGraph CentrePoint Insight Watch) on the non-dominant wrist for the 11-day study period (all day and all night).
4. Take pictures of all of food and drinks consumed, at the start and end (showing food and drink not eaten) of all eating occasions. Participants will use their phones to upload photos to a study website for the entire 11-day study period. Participants will also complete 24-hour dietary recall phone calls for 3 of the 11 study days (i.e., for 1 morning PA day, 1 late afternoon/evening PA day, and 1 no PA day, with the days randomly selected).
5. Complete electronic REDCap surveys, including daily surveys that assess: when (i.e., the exact times) they started eating breakfast, lunch, and dinner that day; when (e.g., the exact times) they went to bed and fell asleep for the night and woke up and got out of bed the next morning, and questions on the quality of their sleep; adverse events and issues with the study equipment (e.g., CGM); and mood state following PA (on days assigned 30 minutes of walking/stepping).

ELIGIBILITY:
Eligibility Criteria

* Singleton, viable pregnancy with low suspicion for clinically significant abnormality or aneuploidy
* Age 18-40 years (at recruitment)
* Comfortable communicating with study staff in English and completing study surveys in English (i.e., no translator needed)
* Identified as Gestational Glucose Intolerance (GGI) and a 3-hr 100g OGTT for Gestational Diabetes Mellitus (GDM) performed ≥ 24 weeks (i.e., GGI or GDM), or GDM by the one step procedure or a 1-hr 50-g glucose challenge test (GCT) ≥ 180 mg/dl performed ≥ 24 weeks

Identification of GGI 1-hr 50-g GCT (non-fasting), with plasma glucose at 1-hr ≥ 130 mg/dL

Identification of GDM by the two-step procedure

Identified as GGI, followed by a 3-hr 100g OGTT at ≥ 24 weeks after an overnight fast, with at least two of four plasma glucose values meeting or exceeding:

* Fasting: 95 mg/dL
* 1-hr: 180 mg/dL
* 2-hr: 155 mg/dL
* 3-hr: 140 mg/dl

Identification of GDM by the one-step procedure 75-g OGTT at ≥ 24 weeks after an overnight fast, with at least one plasma glucose value meeting or exceeding:

* Fasting: 92 mg/dL
* 1-hr: 180 mg/dL
* 2-hr: 153 mg/dL

Identification of GDM by 1-hr 50-g GCT

1-hr 50-g GLT (non-fasting), with plasma glucose at 1-hr ≥ 180 mg/dL at ≥ 24 weeks

Exclusion Criteria

* Indication that physical activity is or should be limited in the current pregnancy
* Previously diagnosed with diabetes (i.e., Type I or Type II diabetes) outside of pregnancy
* Current use of daily medications known to alter insulin resistance and/or metabolic profiles (e.g., metformin, corticosteroids, anti-psychotics)
* Current use of medication for polycystic ovarian syndrome (PCOS) (i.e., history of PCOS okay as long as she is not currently taking medication for PCOS)
* Condition or circumstance that would preclude their ability to follow a strict, time-based study protocol (e.g., psychiatric illness).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CGM glucose outcomes | Throughout the 11-day study period
  Glucose outcome measures include: 24-hour glucose and coefficient of variation, daytime glucose, nighttime glucose, pre-breakfast area under the glucose curve (AUC; calculated for the 120 minutes prior to the start of breakfast), and all post-meal AUCs (calculated for the 120 minutes after the start of the breakfast, lunch and dinner).

SECONDARY OUTCOMES:
Duration of sleep | Throughout the 11-day study period
  Self-reported length of each sleep period (in hours: minutes)
Sleep efficiency | Throughout the 11-day study period
  Self-reported percentage of time spent asleep while in bed (0-100%), for each sleep period
Sleep quality | Throughout the 11-day study period
  Self-reported quality of sleep (i.e., very poor, poor, fair, good, or very good), for each sleep period
Mood | Throughout the 11-day study period (i.e., on days assigned to physical activity)
  Mood following physical activity, using the short version of the Multi-Dimensional Mood Questionnaire (MDMQ, with 15 items) which measures self-reported mood states (i.e., scores range from 15-90, with higher scores indicating better mood state).

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Ehrlich, PhD, Principal Investigator — The University of Tennessee, Knoxville
Locations (1):
- The University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes: all IPD that underlie published results and related data dictionaries available.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available starting 6 months after publication and be available for 3 years.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact Dr. Samantha Ehrlich at sehrlic1@utk.edu

REFERENCES:
- [Derived] Ehrlich SF, Hallenbeck BR, Lewis J, Yousefi F, Miller JI, Zite NB, Fortner KB, Schoutko WW, Crouter SE, Raynor H, Maples JM. Rationale and protocol for the Time to Move Randomized Crossover Trial: morning versus evening time physical activity and CGM-assessed glucose levels in individuals with pregnancy hyperglycemia. Front Clin Diabetes Healthc. 2026 Jan 13;6:1709683. doi: 10.3389/fcdhc.2025.1709683. eCollection 2025. PMID 41607684
- [Derived] Ehrlich SF, Hallenbeck BR, Zite NB, Fortner KB, Paudel A, Raynor HA, Crouter SE, Maples JM. A Randomized Controlled Pilot Trial of a Behavioral Physical Activity Intervention for Pregnancy Hyperglycemia. J Pregnancy. 2025 Nov 20;2025:7485092. doi: 10.1155/jp/7485092. eCollection 2025. PMID 41321483